CLINICAL TRIAL: NCT00700934
Title: Management of Patients With Alpha-1 Antitrypsin Deficiency Associated Emphysema. A National Registry.
Brief Title: Management of Patients With Alpha-1 Antitrypsin Deficiency Associated Emphysema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Docteur Gabriel Thabut, Assistance Publique Hopitaux de Paris
Other Study IDs: 001
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2008-06

CONDITIONS: Alpha 1-Antitrypsin Deficiency; Emphysema
Keywords: FEV1; mortality; Quality of life
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe the natural history of patients with alpha-1 antitrypsin associated emphysema and to figure out associated prognostic factors.

DETAILED DESCRIPTION:
All patients who suffer from this disease are followed every 6 months during a 5 years period. FEV1 decline is the primary endpoint. Quality of life assessed using the Saint George's Respiratory Questionary is recorded too.

ELIGIBILITY:
Inclusion Criteria:

* Serum alpha one antitrypsin < 0.8 g/l
* Emphysema diagnosed by CT scan
* Adult
* Obstructive disorder

Exclusion Criteria:

* Liver or lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emphysema associated alpha-1 antitrypsin deficiency
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-02; Primary Completion 2011-02 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Thabut, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Departement d'épidémiologie, Hôpital Bichat, Paris, France

REFERENCES:
- [Derived] Gauvain C, Mornex JF, Pison C, Cuvelier A, Balduyck M, Pujazon MC, Fournier M, AitIlalne B, Thabut G. Health-related quality of life in patients with alpha-1 antitrypsin deficiency: the French experience. COPD. 2015 May;12 Suppl 1:46-51. doi: 10.3109/15412555.2015.1022645. PMID 25938292
- [Derived] Thabut G, Mornex JF, Pison C, Cuvelier A, Balduyck M, Pujazon MC, Fournier M, AitIlalne B, Porcher R. Performance of the BODE index in patients with alpha1-antitrypsin deficiency-related COPD. Eur Respir J. 2014 Jul;44(1):78-86. doi: 10.1183/09031936.00168113. Epub 2014 Feb 13. PMID 24525449